CLINICAL TRIAL: NCT05740748
Title: A Phase 2 Multi-centre Randomized Double-blind Placebo-controlled Parallel Group Study to Examine the Effects of 24 Weeks Tezepelumab 210 mg sc q4wks on Methacholine Airway Hyperresponsiveness in Participants With Mild Allergic Asthma
Brief Title: Tezepelumab and Methacholine Airway Hyperresponsiveness in Participants With Mild Allergic Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESR-22-21828
Record Dates: First submitted 2023-02-06; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Asthma, Allergic
Keywords: asthma; airway hyperresponsiveness; mast cell; Thymic stromal lymphopoietin; tezepelumab
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tezepelumab (Experimental): tezepelumab 210 mg sc q4wks 20 weeks treatment
  Interventions: Drug: Tezepelumab
- Placebo (Placebo Comparator): placebo sc q4wks 20 weeks treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tezepelumab — tezepelumab 210 mg sc q4wks for 20 weeks
  Arms: Tezepelumab
Drug: Placebo — placebo sc q4wks for 20 weeks
  Arms: Placebo

SUMMARY:
Asthma is a condition where small inhaled particles can cause inflammation in the lung leading to constriction of airways and wheeze. Mast cells are immune cells in airways that can release chemical causing constriction of the airways and wheeze. Tezepelumab is an injectable medication that improves asthma by stopping inflammation, but the effect on mast cells is not known. Tezepelumab was approved in Canada July 2022 for treatment of severe asthma. Tezepelumab is not approved for treatment of mild asthma by any health authority, except for use in research studies like this. This study will examine the effect of tezepelumab on mast cells and airway constriction to understand the mechanisms of asthma, and which patients will benefit most from drugs like tezepelumab.

DETAILED DESCRIPTION:
The proposed study will address whether tezepelumab has the unique ability to improve AHR in participants with mild allergic asthma.

This is a phase 2 multi-centre randomized double-blind placebo-controlled parallel-group study to examine the effects of 24 weeks tezepelumab 210 mg sc q4wks on methacholine airway hyperresponsiveness in participants with mild allergic asthma, stratified for sex and sensitivity to seasonal allergens.

There are 9 study visits over a period of 27 weeks (Figure 1). Study procedures performed at Weeks -1, 8, 16 and 24 will be divided across 2 visits at least 48 hours apart for measurement of AHR to methacholine first, and mannitol at least 48 hours later.

The screening period at Week -1 will determine eligibility. At Week -1, eligible allergic mild asthmatic participants will be randomized 1:1 to placebo or tezepelumab 210 mg subcutaneous administered monthly for a total of 24 weeks. AHR will be measured by methacholine and mannitol challenges at baseline (Week -1) performed at least 48 hours apart. Changes in AHR response will be measured by repeat methacholine and mannitol challenges at Weeks 8, 16 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male and female 18 through 65 years of age
3. Positive skin-prick test to a common aeroallergen
4. Methacholine PD20 ≤ 200mcg
5. Mannitol DRR ≤ 42.3mg/FEV1 %f all (equivalent to PD15 ≤ 635mg)
6. Baseline FEV1 ≥ 70% of the predicted value
7. Negative pregnancy test (urine) for female participants of childbearing potential.

Exclusion Criteria:

1. Current or former smoker with >10-pack-year history
2. Current or previous history of lung disease other than mild stable allergic asthma
3. Significant systemic disease, including history of current malignancy or autoimmune disease
4. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
5. Previous randomisation in the present study. Re-screening (Week -1) for FEV1 and AHR is permitted once for each test.
6. Participation in another clinical study with an investigational product during the last 30 days or 5 half-lives of the drug (whichever is longer)
7. Use of any medications for treatment of asthma other than prophylactic short-acting β2-agonists, or use of short-acting β2-agonists for relief of symptoms less than once weekly.
8. Participants with known hypersensitivity to tezepelumab or any of the excipients of the product.
9. Positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening
10. Known to have tested positive for human immunodeficiency virus
11. Known history of drug or alcohol abuse within 1 year of screening
12. For women only - currently pregnant (confirmed with positive pregnancy test) or breast feeding.
13. Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Methacholine PD20 | Week -1 to Week 24
  The provocative dose of methacholine causing 20% fall in FEV1

SECONDARY OUTCOMES:
Dose response ratio to mannitol | Week -1 to Week 24
  The mannitol dose response ratio calculated by dividing the total cumulative dose by the % fall in FEV1 at that dose.
Mast cell tryptase levels. | Week -1 to Week 24
  Level of mast cell-derived tryptase in blood and urine at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No